CLINICAL TRIAL: NCT06918470
Title: Research on the Effect of Noise Cancelling Headphones in Reducing Postoperative Pain During Gynecological Laparoscopic Surgery ：a Randomized Controlled Trial
Brief Title: Research on the Effect of Noise Cancelling Headphones in Reducing Postoperative Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maternal and Child Health Hospital of Hubei Province (Other)
Responsible Party: Principal Investigator, Li Na, Deputy Chief Physician, Maternal and Child Health Hospital of Hubei Province
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCHH_011
Record Dates: First submitted 2025-03-28; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Noise Cancelling Headphones; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional processing group, (Sham Comparator): Standard monitoring techniques ,Conventional processing without noise cancelling headphones
  Interventions: Other: Standard monitoring techniques
- wearing noise cancelling headphones group (Experimental): group started wearing noise cancelling headphones until the end of the surgery in the general anesthesia induction group to isolate intraoperative environmental noise
  Interventions: Other: noise cancelling headphones

INTERVENTIONS:
Other: Standard monitoring techniques — （3）atients were given the same anesthesia regimen. Standard monitoring techniques include electrocardiogram, pulse oximeter, heart rate and blood pressure monitoring, continuous monitoring of bispecific index of electroencephalography, and the use of remifentanil (0.3 mg/kg) Rapid sequence induction was performed using sufentanil (0.3 μ g/kg), propofol (2.5mg/kg), and rocuronium bromide (0.6 mg/kg). Anesthesia was maintained using remifentanil (0.1-0.2 μ g/0kg/min), inhaled sevoflurane (1%), and intravenous propofol (1-4 mg/kg/h) to maintain BIS 40-60, with heart rate and blood pressure within 20% of baseline values.
  Arms: Conventional processing group,
Other: noise cancelling headphones — The treatment group started wearing noise cancelling headphones until the end of the surgery in the general anesthesia induction group to isolate intraoperative environmental noise,patients were given the same anesthesia regimen. Standard monitoring techniques include electrocardiogram, pulse oximeter, heart rate and blood pressure monitoring, continuous monitoring of bispecific index of electroencephalography, and the use of remifentanil (0.3 mg/kg) Rapid sequence induction was performed using sufentanil (0.3 μ g/kg), propofol (2.5mg/kg), and rocuronium bromide (0.6 mg/kg). Anesthesia was maintained using remifentanil (0.1-0.2 μ g/0kg/min), inhaled sevoflurane (1%), and intravenous propofol (1-4 mg/kg/h) to maintain BIS 40-60, with heart rate and blood pressure within 20% of baseline values.
  Arms: wearing noise cancelling headphones group

SUMMARY:
this randomized controlled trial selects patients undergoing gynecological laparoscopy under general anesthesia. By using noise reduction earphones during surgery, the patient's postoperative pain score and demand for opioids are observed, providing a basis and reference for the efficacy and safety of noise reduction earphones in gynecological endoscopic surgery.

DETAILED DESCRIPTION:
Every year, 200 million surgical procedures are performed worldwide, and 40-65% of patients experience moderate to severe pain after surgery Failure to provide sufficient postoperative analgesia increases the risk of surgical complications and affects patients' early activity and recovery . Opioids are still the main method of treatment, and their side effects include urinary retention, itching, nausea, vomiting, postoperative intestinal obstruction, dizziness and cognitive impairment . Researchers pay more and more attention to non pharmacology and non-invasive analgesia methods, including music therapy, traditional Chinese medicine acupuncture and moxibustion and watching educational videos . Due to the introduction of various surgical tools, the noise pollution in the operating room has gradually intensified, affecting surgical patients and medical staff. Previous studies have shown that general anesthesia does not hinder the brain's processing ability for sound and language; The patient's auditory cortex remains active , and even in anesthesia induced coma, the patient can still maintain the ability to understand auditory information. Other recent studies have found that intraoperative exposure to positive auditory stimuli, including music, treatment suggestions and white noise, can reduce postoperative pain, environmental protection, and acupuncture and moxibustion can also have a similar positive impact . Therefore, this randomized controlled trial selects patients undergoing gynecological laparoscopy under general anesthesia. By using noise reduction earphones during surgery, the patient's postoperative pain score and demand for opioids are observed, providing a basis and reference for the efficacy and safety of noise reduction earphones in gynecological endoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

ASA grade I or II, aged 18-55 years , female were selected for gynecological laparoscopy under elective general anesthesia. -

Exclusion Criteria:

History of serious illness requiring further care in the intensive care unit after surgery; Abnormal hearing; Postoperative mechanical ventilation or continued anesthesia or sedation is required; Preoperative chronic pain or long-term use of painkillers; other factors that hinder patients from cooperating with the research plan

-

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-05-12 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
pain scores | 6, 12, and 24 hours postoperatively
  the patient's resting and exercise induced pain scores,by the Visual Analog Scale (VAS) It typically involves a 10-centimeter horizontal or vertical line, with endpoints labeled "no pain" (0) and "worst pain imaginable" (10).
maximum pain scores | at 0-6 hours, 6-12 hours, and 12-24 hours postoperatively.
  maximum pain scores at 0-6 hours, 6-12 hours, and 12-24 hours postoperatively.by the Visual Analog Scale (VAS) It typically involves a 10-centimeter horizontal or vertical line, with endpoints labeled "no pain" (0) and "worst pain imaginable" (10).

SECONDARY OUTCOMES:
maximum resting pain score | within 24 hours postoperatively
  by the Visual Analog Scale (VAS) It typically involves a 10-centimeter horizontal or vertical line, with endpoints labeled "no pain" (0) and "worst pain imaginable" (10).
total opioid consumption | within 24 hours postoperatively
the number of PCIA pump buttons | within 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Na Li, MD, Principal Investigator — Maternal and Child Health Hospital of Hubei Province
Locations (1):
- Maternal and Child Health Hospital of Hubei Province,, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No